CLINICAL TRIAL: NCT01412645
Title: Long-term Investigation of Resveratrol on Management of Metabolic Syndrome, Osteoporosis and Inflammation, and Identification of Plant Derived Anti-inflammatory Compounds
Brief Title: Long-term Investigation of Resveratrol in Obesity
Acronym: LIRMOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LIRMOI
Record Dates: First submitted 2011-07-13; First posted 2011-08-09 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Inflammation; Insulin Sensitivity; Osteoporosis
Keywords: Obesity; Inflammation; Metabolic Syndrome; Insulin sensitivity; Osteoporosis; Bone turnover; Ectopic fat accumulation; Resveratrol
MeSH Terms: conditions — Obesity; Inflammation; Insulin Resistance; Osteoporosis; Metabolic Syndrome | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Resveratrol
- High-dose Resveratrol (Experimental)
  Interventions: Dietary Supplement: Resveratrol
- Low-dose Resveratrol (Experimental)
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — 500mg resveratrol 2 times daily for 4 months (High-dose Resveratrol), 75mg resveratrol 2 times daily for 4 months (Low-dose Resveratrol) or
  1 placebo 2 times daily for 4 months

SUMMARY:
The aim of this study is to investigate potential metabolic effects of resveratrol in men with metabolic syndrome(otherwise healthy).

The investigators hypothesize that resveratrol has an anti-inflammatory effect, and will increase insulin sensitivity, change the fat- and sugar-metabolism, and down-regulate bone-turnover.

DETAILED DESCRIPTION:
The study will be done in a collaboration between two PhD students, who focus on effects in adipose- and muscle- tissue, and bone tissue respectively.

The investigators will look at changes in

* inflammation-markers
* biochemical markers of fat- and sugar-metabolism
* gene-expression in fat- and muscle-tissue
* body composition (DXA (whole body) and MR spectroscopy)
* biochemical markers of bone-metabolism
* Bone Mineral Density (DXA scans)
* bone structure (QCT)
* gene-expression and cytokines in bone marrow

Some of the volunteers will have their insulin sensitivity measured.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 30-60 years old
* Metabolic Syndrome
* Written informed consent

Exclusion Criteria:

* Diabetes, thyroid or parathyroid disease, hypogonadism
* Treatment-requiring osteoporosis
* Heart, liver or kidney disease
* Present or previous malignancy
* MR contraindication
* Alcohol dependency
* Weight > 130 kilograms

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in markers of inflammation (hs-CRP) in blood after 4 months of treatment with either resveratrol or placebo | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Steen B Pedersen, MD, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Clinical Institute, Aarhus University, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Kjaer TN, Ornstrup MJ, Poulsen MM, Stodkilde-Jorgensen H, Jessen N, Jorgensen JOL, Richelsen B, Pedersen SB. No Beneficial Effects of Resveratrol on the Metabolic Syndrome: A Randomized Placebo-Controlled Clinical Trial. J Clin Endocrinol Metab. 2017 May 1;102(5):1642-1651. doi: 10.1210/jc.2016-2160. PMID 28182820
- [Derived] Ornstrup MJ, Harslof T, Kjaer TN, Langdahl BL, Pedersen SB. Resveratrol increases bone mineral density and bone alkaline phosphatase in obese men: a randomized placebo-controlled trial. J Clin Endocrinol Metab. 2014 Dec;99(12):4720-9. doi: 10.1210/jc.2014-2799. PMID 25322274